CLINICAL TRIAL: NCT02410577
Title: A Pilot Study of 89Zr-J591 Anti-Prostate-Specific Membrane Antigen Monoclonal Antibody in Patients With Glioblastoma Multiforme
Brief Title: 89Zr-J591 Anti-Prostate-Specific Membrane Antigen Monoclonal Antibody in Patients With Glioblastoma Multiforme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-002
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-08

CONDITIONS: Glioblastoma
Keywords: 89Zr-J591; 15-002
MeSH Terms: conditions — Glioblastoma | interventions — Positron Emission Tomography Computed Tomography; Blood Specimen Collection

ARMS (1):
- 89Zr-J591 (Experimental): Patients will not be required to fast prior to imaging with 89Zr-J591 injection or imaging. The total dose of humanized mAb J591 will be 20mg. Patients will first receive an injection of 18-19mg of unchelated J591 to reach the total administered dose of antibody (IND11407) followed by 5 mCi (+/- 10%) of 89Zr-J591 (1 to 2 mg). Administration of the cold antibody will be followed by the labeled compound.
  Interventions: Drug: 89Zr-J591; Device: PET/CT Scan; Device: MRI; Other: Blood draw

INTERVENTIONS:
Drug: 89Zr-J591 — The intervention is the administration of an injection of 18-19mg of unchelated J591 to reach the total administered dose of antibody followed by 5 mCi (+/- 10%) of 89Zr-J591 (1 to 2 mg) . After administration of the experimental tracer, the patient will undergo a Brain PET/CT scan 24 hours, 48 hours post injection and 3-8 days. The 48 hour scan is strongly suggested, but optional.
Device: PET/CT Scan
Device: MRI
Other: Blood draw — Bloods samples will be drawn immediately before and approximately 30 minutes after 89Zr-J591 injection.

SUMMARY:
The purpose of this study is to test a new imaging agent called 89Zr-J591 (stands for humanized antibody called J591, that is attached to a radioactive material called Zirconium-89) in patients with glioblastoma multiforme.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 25 years old and < 80 years old
* Patients with reoccurrence of brain tumor
* The principal investigator or co-PI must review MRI and CT findings based on the radiologic assessment provided they meet the following imaging criteria (as established in the clinical trial 09-177):

OR

* Patients with newly diagnosed GBM and one of the following options:
* Eligible for surgery after the last research scan.
* Significant residual disease after initial surgery
* The principal investigator or co-PI must review MRI and CT findings and agree with the presence of significant residual disease
* Treatment (non-surgical) naïve
* Karnofsky Performance Score ≥ 70

Exclusion Criteria:

* Laboratory values:

  * Serum creatinine >2.5 mg/dL.
  * AST (SGOT) >2.5x ULN.
  * Bilirubin (total) >1.5x ULN.
  * Serum calcium >11 mg/dL.
* Pregnant or breastfeeding (if a female is of childbearing potential, and unsure of pregnancy status, a standard pregnancy test should be done).
* If an initial biopsy demonstrates neoplasm other than GBM
* Presence of any other co-existing condition which, in the judgment of the investigator, might increase the risk to the subject.
* Presence of serious systemic illness, including: uncontrolled inter-current infection, uncontrolled malignancy, significant renal disease, or psychiatric/social situations, which might limit compliance with study requirements
* Prior treatment.
* Other serious illness (es), which might preclude completion of this, study or interfere with determination of causality of any adverse effects experienced in this study.

Ages: 26 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Osborne, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] McBriar JD, Shafiian N, Scharf S, Boockvar JA, Wernicke AG. Prostate-Specific Membrane Antigen Use in Glioma Management: Past, Present, and Future. Clin Nucl Med. 2024 Sep 1;49(9):806-816. doi: 10.1097/RLU.0000000000005365. Epub 2024 Jul 1. PMID 38968568
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- 89Zr-J591: Patients will not be required to fast prior to imaging with 89Zr-J591 injection or imaging. The total dose of humanized mAb J591 will be 20mg. Patients will first receive an injection of 18-19mg of unchelated J591 to reach the total administered dose of antibody (IND11407) followed by 5 mCi (+/- 10%) of 89Zr-J591 (1 to 2 mg). Administration of the cold antibody will be followed by the labeled compound.
  89Zr-J591: The intervention is the administration of an injection of 18-19mg of unchelated J591 to reach the total administered dose of antibody followed by 5 mCi (+/- 10%) of 89Zr-J591 (1 to 2 mg) . After administration of the experimental tracer, the patient will undergo a Brain PET/CT scan 24 hours, 48 hours post injection and 3-8 days. The 48 hour scan is strongly suggested, but optional.
  PET/CT Scan
  MRI
  Blood draw: Bloods samples will be drawn immediately before and approximately 30 minutes after 89Zr-J591 injection.
Period: Overall Study
Arm/Group | 89Zr-J591
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 89Zr-J591
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 56 [51 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Binding of 89Zr-J591
Description: This will be measured by J591 uptake in PET scan.
Time Frame: 1 year
Population: Data were not collected.
Arm/Group | 89Zr-J591
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | 89Zr-J591
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT02410577/Prot_SAP_000.pdf